CLINICAL TRIAL: NCT01926925
Title: Endothelial Function in Hispanic Children/Adolescents at Risk for Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Joslin Diabetes Center (Other)
Responsible Party: Principal Investigator, Enrique Caballero, Clinical Investigator/Director Latino Diabetes Initiative, Joslin Diabetes Center
Other Study IDs: CHS#: 01-14
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Obesity; Insulin Resistance
Keywords: Type 2 diabetes, Endothelium, children/adolescents
MeSH Terms: conditions — Obesity; Insulin Resistance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Overweight Hispanic children/adolescents
- 2: Lean Hispanic children/adolescents

SUMMARY:
Type 2 diabetes is now more frequent in children/adolescents, especially in those from minority populations, including Hispanic Americans (HA). Diabetes and the pre-diabetes state markedly increase the risk of cardiovascular disease. Endothelial dysfunction is seen in the earliest stages of atherogenesis, which ultimately leads to cardiovascular disease. The main aim of this study is to evaluate the endothelial function in HA children/adolescents who are at risk for developing type 2 diabetes (obese children/adolescents from the Hispanic population).

The investigators' hypothesis is that endothelial dysfunction is present in this population and that it is associated with metabolic abnormalities linked to the insulin resistance syndrome. The investigators will study 2 groups of 15 individuals each, age 10-18 years. Group 1 will consist of obese (body mass index greater than 85th percentile for age and sex) Hispanic American children/adolescents and group 2 will consist of healthy, non-overweight (body mass index between the 25th and 50 th percentile for age and sex) Hispanic American children/adolescents.

The study will be carried out at the Joslin Diabetes Center. During the first day, participants will have a medical history and full physical examination, a standard OGTT and measurement of blood cell count, plasma glucose, insulin, lipids, HbA1c, BUN, creatinine, electrolytes, estradiol, testosterone, free fatty acids, CRP, endothelial markers, urinary microalbumin and hCG, if appropriate. An OGTT will be performed in order to rule out IGT or Diabetes. Estimations of insulin secretion and insulin sensitivity will be assessed using the homeostasis model assessment (HOMA). In the second day, the body composition and the brachial artery vasodilatory response to hyperemia will be assessed. Those found with diabetes will be tested for GAD-65 and IA2.

The investigators' hypothesis is that Hispanic American children/adolescents at risk for type 2 diabetes have impaired endothelial function and vascular reactivity that are associated with the degree of insulin resistance and its metabolic abnormalities.

DETAILED DESCRIPTION:
Information as above

ELIGIBILITY:
Inclusion Criteria:

* Group 1:

  1. Age between 10-18 years;
  2. Hispanic (we will consider a subject being Hispanic if both parents are reported as Hispanics when asked the following question: "What ethnic group do you consider that you belong to?");
  3. No history of type 2 diabetes in any first-degree relative;
  4. Body mass index between the 25th and 50th percentile for age and sex
  5. Not have participated in any exercise program for the 6 months prior to the beginning of the study.

Group 2:

1. Age between 10-18 years;
2. Hispanic (same criteria as above);
3. Body mass index greater than the 85th percentile for age and sex;
4. Not have participated in any exercise program for the 6 months prior to the beginning of the study.

Exclusion Criteria:

* The exclusion criteria include: diabetes, pregnancy, smoking, cardiovascular disease, uncontrolled hypertension, renal disease, proteinuria, cancer, infectious diseases, severe GI diseases, lung disease, electrolyte abnormalities, anemia, endocrine disorders, severe dyslipidemia, peripheral vascular disease, medications: beta-blockers, any diuretic, calcium channel blockers, ACE inhibitors, niacin, glucocorticoids, any antineoplastic agent, antibiotics, psychoactive agents, bronchodilators or insulin.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Hispanic children/adolescents
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2001-05; Primary Completion 2010-05 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Plasma levels of markers of endothelial activation and vascular inflammation | cross sectional study - one time evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Caballero, MD, Principal Investigator — Joslin Diabetes Center